CLINICAL TRIAL: NCT01059396
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study on the Effectiveness of Treatment With Beta-blockers to Prevent Decompensation of Cirrhosis With Portal Hypertension
Brief Title: Study on B-blockers to Prevent Decompensation of Cirrhosis With HTPortal
Acronym: PREDESCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PREDESCI
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-01

CONDITIONS: Portal Hypertension Gastropathy; Esophageal Varices; Spontaneous Bacterial Peritonitis; Hepatic Encephalopathy; Ascites
MeSH Terms: conditions — Esophageal and Gastric Varices; Hepatic Encephalopathy; Ascites | interventions — Propranolol; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propranolol (Experimental)
  Interventions: Drug: propranolol
- carvedilol (Experimental)
  Interventions: Drug: carvedilol
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: propranolol — GPVH ≥ 10 mmHg - responders: propranolol.
  Arms: Propranolol
Drug: carvedilol — GPVH ≥ 10 mmHg nonresponders: carvedilol.
  Arms: carvedilol
Drug: placebo — placebo propranolol / carvedilol
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study on the effectiveness of treatment with beta-blockers to prevent decompensation of cirrhosis with portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years old.
* With liver cirrhosis diagnosed by previous biopsy or by clinical criteria, and analytical image.
* No esophageal varices (or with small varices without red signs) in a recent videogastroscophy (<3 months before randomization).
* Absence of ascites demonstrated by a recent ultrasound (<3 months before the randomization).
* informed consent

Exclusion Criteria:

* previous decompensation of liver cirrhosis associated with portal hypertension.
* GPVH <10 mmHg.
* Portal axis thrombosis affecting the portal trunk or main hepatic branches, or the splenic or mesenteric vein.
* Hepatocellular carcinoma demonstrated by two imaging tests.
* Bilirubin> 3 mg / dl (or> 50 micromol / l), platelets <30 x10E9/lo Quick <30%.
* Presence of renal insufficiency (serum creatinine> 2 mg / dl or> 200 micromol / l).
* Any comorbidity involving a therapeutic limitation and / or a prognosis of life <12 months.
* Absolute contraindication to treatment with β-blockers (severe bronchospasm, stenosis aortic A-V block, intermittent claudication, severe psychosis, bronchial asthma)
* Hypersensitivity to β-blockers.
* Pregnancy or lactation.
* To receive anticoagulant treatment.
* Past treatment with nitrated or β-blockers in the two weeks prior inclusion.
* Cirrhosis C virus active antiviral therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2010-01-28 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Appearance of complications of portal hypertension: bleeding (caused by portal hypertension gastropathy and / or esophageal varices), ascites and / or spontaneous bacterial peritonitis(PBE), hepatic encephalopathy. Death from any cause. | 3 years

SECONDARY OUTCOMES:
Compare the appearance of each of the complications of portal hypertension (ascites, SBP and other bacterial infections, varicose veins or signs of high risk, upper gastrointestinal bleeding portal hypertension, hepatic encephalopathy). | 3 years
Assess the development of liver failure. | 3 years
Quantify the adverse effects of treatment (occurrence and intensity, need to withdraw the treatment). | 3 years
To assess survival. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Càndid Villanueva Sánchez, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (8):
- Spain (8):
  - Hospital German Trias i Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de la Vall d'Hebron, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Clínica Puerta del Hierro, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid

REFERENCES:
- [Derived] Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Brujats A, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J; PreDesCI Study Investigators. Bacterial infections adversely influence the risk of decompensation and survival in compensated cirrhosis. J Hepatol. 2021 Sep;75(3):589-599. doi: 10.1016/j.jhep.2021.04.022. Epub 2021 Apr 24. PMID 33905794
- [Derived] Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J. beta blockers to prevent decompensation of cirrhosis in patients with clinically significant portal hypertension (PREDESCI): a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2019 Apr 20;393(10181):1597-1608. doi: 10.1016/S0140-6736(18)31875-0. Epub 2019 Mar 22. PMID 30910320